CLINICAL TRIAL: NCT01018017
Title: A Phase IIa, Randomized, Placebo-Controlled, Double-Blind Clinical Study to Assess the Safety, Tolerability, and Activity of Oral SRT2104 Capsules Administered for 28 Days to Subjects With Type 2 Diabetes Mellitus
Brief Title: A Clinical Study to Assess the Safety, Tolerability, and Activity of Oral SRT2104 Capsules Administered for 28 Days to Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 114010
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SRT2104

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2.0g SRT2104 (Active Comparator): The 2.0g SRT2104 treatment group will be administered eight SRT2104 capsules per day. 2.0g SRT2104 will be administered orally once daily for twenty-eight consecutive days. During non-clinic days, the subject will self-administer the test material approximately 15 minutes following consumption of a standard morning meal at home (200 cc of Ensure Plus®).
  Interventions: Drug: SRT2104
- Placebo (Placebo Comparator): The placebo treatment group will be administered eight placebo capsules per day. Placebo will be administered orally once daily for twenty-eight consecutive days. During non-clinic days, the subject will self-administer the test material approximately 15 minutes following consumption of a standard morning meal at home (200 cc of Ensure Plus®).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — For placebo product, the SRT2104 drug substance will be replaced by microcrystalline cellulose (Avicel® PH 105) to match the SRT2104 investigational product.
  Arms: Placebo
Drug: SRT2104 — SRT2104 will be supplied as hard gelatin capsules, with each containing 250mg SRT2104.
  Arms: 2.0g SRT2104

SUMMARY:
Randomized, placebo-controlled, parallel-group, double-blind, multiple-dose, activity and safety clinical study of SRT2104 administered orally once daily for 28 consecutive days. This will be an inpatient/outpatient study to assess the safety and pharmacokinetics of SRT2104 in type 2 diabetic male and female subjects on an existing, stable, background metformin therapy. Approximately 80 subjects will be enrolled. Subjects will be evenly randomized to receive SRT2104 2.0 g/day or placebo in the fed state.

Subjects will be required to stay overnight at the study center on Days -2, -1, 0, 1 (optional discharge at investigator's discretion), 27, 28, 41, and 42. During these admissions, pharmacokinetic, biomarker and glycated albumin samples will be collected, and glucose profiling, OGTT, glucose stabilization, hyperinsulinemc euglycemic clamp (HEGC) studies with indirect calorimetry and various other safety and activity procedures will be performed. On Day 1 of the study, subjects will be randomized to receive SRT2104 or placebo. Day 43 will be the last day of the study and subjects will be released. In addition, subjects will be asked to return to the study center on Day 14 for interim safety assessments.

During the dosing period, study personnel will contact subjects by telephone on Days 7 and 21 to conduct a safety assessment. Subjects will be required to monitor their fasting blood glucose and complete a daily diary for the outpatient portion of the study between Days 1 and 28. A follow-up, safety phone call will occur 30 days following their final dose of SRT2104 or placebo (Day 58 of the study) to identify any possible additional adverse events or concomitant medications.

DETAILED DESCRIPTION:
Randomized, placebo-controlled, parallel-group, double-blind, multiple-dose, activity and safety clinical study of SRT2104 administered orally once daily for 28 consecutive days. This will be an inpatient/outpatient study to assess the safety and pharmacokinetics (PK) of SRT2104 in type 2 diabetic (T2D) male and female subjects on an existing, stable, background metformin therapy. Approximately 112 subjects aged 18-65 years, who fulfill the inclusion/exclusion criteria, will be screened for this study to enroll approximately 80 subjects. Subjects will be evenly randomized to receive SRT2104 2.0 g/day or placebo approximately 15 minutes following consumption of a standardized morning meal. Subjects will remain on a fixed dose of test material for all dosing days in the study.

Subjects will sign the informed consent form at the Screening Visit, and will undergo screening assessments to verify eligibility for the study. If eligible and willing to participate, subjects will return to the clinic within 21 days of the Screening Visit to participate in the pre-dosing phase of the study. On Day 1 of the study, subjects will be randomized to receive SRT2104 or placebo. Subjects will be required to stay overnight at the study center on Days -2, -1, 0, 1 (optional discharge at investigator's discretion), 27, 28, 41, and 42 for testing, to assess safety, and to gather required biomarker samples. In addition, subjects will be asked to return to the study center on Day 14 for interim safety assessments. The subject will be telephoned on Days 7 and 21 to assess safety. Subjects will be required to monitor their fasting blood glucose and complete a daily diary for the outpatient portion of the study between Days 1 and 28. A follow-up, safety phone call will occur 30 days following their final dose of SRT2104 or placebo (Day 58 of the study) to identify any possible additional adverse events (AEs) or concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent to participate in the study
* Ambulatory male and female subjects (of any race) with T2D within the age range of 18-65 years (inclusive) at the time of screening
* All female subjects must be of non-childbearing potential. All male subjects must agree with their partners to use double-barrier birth control or abstinence while participating in the study and for 12 weeks following the last dose of investigational product. For the purposes of this study, non-childbearing is defined as:

  * Amenorrheic for at least 12 consecutive months; menopausal status in amenorrheic females will be confirmed by demonstrating levels of follicle stimulating hormone (FSH) >40-138 mIU/mL and estradiol < 30 pg/mL at entry. In the event a subject's menopause status has been clearly established (for example, the subject indicates she has been amenorrheic for 10 years), but FSH and/or estradiol levels are not consistent with a post-menopausal condition, determination of subject eligibility will be at the discretion of the principal investigator with agreement of the independent medical monitor
  * At least 6 weeks post-surgical bilateral oophorectomy (with or without hysterectomy) or post tubal ligation
* The subject must be on stable metformin monotherapy for a minimum of 3 months prior to the Screening visit.
* HbA1c of 6.5%-9.5% (inclusive)
* Body Mass Index (BMI) of 22-38 kg/m^2 (inclusive)
* Resting supine blood pressure (BP) < 160/90 mmHg
* Have a normal 12-lead electrocardiogram (ECG) or one with changes considered to be clinically insignificant on medical review and QTc intervals as defined below:

  * QTcB must be <450 msec for males and <470 msec for females (based on single or average QTc value of triplicate ECGs obtained over a brief period)
  * QTcB must be <480 msec in subjects with Bundle Branch Block
* Comprehension of the nature and purpose of the study and able to comply with the protocol requirements
* Able to communicate in person and by telephone in a manner that allows all protocol procedures to be carried out safely and reliably in the opinion of the investigative site staff

Exclusion Criteria:

* Any major illness in the 3 months prior to study entry or any significant ongoing chronic medical illness not related to diabetes (e.g., recent myocardial infarction, unstable angina, stroke, or transient ischemic attack) which in the opinion of the principal investigator or medical monitor could risk subject safety or interpretation of the results
* Renal or liver impairment, defined as:

  * Serum creatinine level of ≥ 1.4 mg/dL for females and ≥ 1.5 mg/dL for males
  * AST and ALT ≥ 2xULN
  * alkaline phosphatase and bilirubin > 1.5xULN (an isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%)
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of Screening
* A positive test for HIV antibody
* History of or current gastrointestinal diseases influencing drug absorption as judged by the investigator
* Significant history of alcoholism or drug/chemical abuse, or a positive result of the urine drug/alcohol screen at the Screening Visit, or consuming more than 28 units of alcohol per week (one unit of alcohol equals about 250 mL of beer or lager, one glass of wine, or 20 mL spirits)
* Participation in any clinical trial within 3 months prior to the first dose of investigational product in the current study
* History of difficulty in donating blood or accessibility of veins in left or right arm
* Donation or loss of blood (more than 500 mL) within 3 months prior to receiving the first dose of investigational product
* Use of any prescription drug therapy, with the exception of any prescription medication administered at a stable dose for at least 6 weeks prior to Screening, provided the medication is not contraindicated by the metformin label (see Appendix A for Glucophage® Summary of Product Characteristics)
* Use of any anti-diabetic therapy other than metformin, within 3 months of the first dose of investigational product
* Use of any dietary or herbal supplements within 3 weeks prior to the first dose of investigational product
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation
* Active neoplastic disease or history of neoplastic disease within 5 years of study entry (except for basal cell carcinoma of the skin or carcinoma in situ)
* Increased risk of thrombosis, e.g., subjects with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-03-03 (Actual); Primary Completion 2010-12-25 (Actual); Study Completion 2010-12-25 (Actual)

PRIMARY OUTCOMES:
The areas under the glucose concentration time curve from time 0 (dosing) to 2 hours post-dose (AUC 0-2h, glucose) obtained during an oral glucose tolerance test (OGTT) on days 28 and 42. | Day 28 and Day 42
  AUC 0-2h, glucose was obtained pre-dose (Day -1), at the end of the dosing period (Day 28), and at end-of-study (Day 42). Blood samples were obtained prior to administration of 75 g of oral glucose which was administered as standard glucose beverage after an overnight fast, within 15 minutes. A peripheral blood sample was drawn from a peripheral arm vein prior to the participant consuming the beverage. Additional blood samples were drawn at 30, 60, 90, and 120 minutes after the participant had consumed the glucose beverage for the measurement of glucose, insulin and C-peptide concentrations. Blood glucose concentrations were determined with a glucose analyzer. On Day 28, on which the participant received also investigational product, the OGTT had to be performed prior to consumption of standard meal and administration of investigational product.
The areas under the serum insulin concentration time curve from time 0 (dosing) to 2 hours post-dose (AUC 0-2h, insulin) obtained during OGTT, on days 28 and 42. | Day 28 and 42
  AUC 0-2h, insulin was obtained pre-dose (Day -1), at the end of the dosing period (Day 28), and at end-of-study (Day 42). Blood samples were obtained prior to administration of 75 g of oral glucose which was administered as standard glucose beverage after an overnight fast, within 15 minutes. A peripheral blood sample was drawn from a peripheral arm vein prior to the participant consuming the beverage. Additional blood samples were drawn at 30, 60, 90, and 120 minutes after the participant had consumed the glucose beverage for the measurement of glucose, insulin and C-peptide concentrations. Blood glucose concentrations were determined with a glucose analyzer. On Day 28, on which the participant received also investigational product, the OGTT had to be performed prior to consumption of standard meal and administration of investigational product.unit of measurement was microunits×hours per milliliter
Measurement of insulin sensitivity consisting of the insulin sensitivity index (ISIest) obtained during OGTT. | Up to Day 42
  Stumvoll Index: ISIest was obtained pre-dose (Day -1), at the end of the dosing period (Day 28), and at end-of-study (Day 42). Blood samples were obtained prior to administration of 75 g of oral glucose which was administered as standard glucose beverage after an overnight fast, within 15 minutes. ISI is based on insulin and glucose levels in a fasting state during OGTT and is calculated as: ISI (Matsuda) = 10000/√ G0 X I0 X Gmean X Imean where G0 - fasting plasma glucose (mg/dL) I0 - fasting plasma insulin (milliinternational units (miU)/L) Gmean - mean plasma glucose during OGTT (mg/dL) Imean - mean plasma insulin during OGTT (mIU/L). Unit of measure was (Deciliter × liter)(mg × milliinternational units)
Measurement of insulin sensitivity consisting of the composite whole body sensitivity index (ISIcomposite) obtained during OGTT | Up to Day 42
  ISI is based on insulin and glucose levels in a fasting state during an oral glucose tolerance test (OGTT) and is calculated as: ISI (Matsuda) = 10000/√ G0 X I0 X Gmean X Imean where G0 - fasting plasma glucose (mg/dL) I0 - fasting plasma insulin (mIU/L) Gmean - mean plasma glucose during OGTT (mg/dL) Imean - mean plasma insulin during OGTT (mIU/L). ISIcomposite was obtained pre-dose (Day -1), at the end of the dosing period (Day 28), and at end-of-study (Day 42).
Measurement of insulin sensitivity consisting of the hepatic insulin sensitivity (HIRI) obtained during OGTT | Up to Day 42
  HIRI was obtained pre-dose (Day -1), at the end of the dosing period (Day 28), and at end-of-study (Day 42). Blood samples were obtained prior to administration of 75 g of oral glucose which was administered as standard glucose beverage after an overnight fast, within 15 minutes. A peripheral blood sample was drawn from a peripheral arm vein prior to the participant consuming the beverage. Additional blood samples were drawn at 30, 60, 90, and 120 minutes after the participant had consumed the glucose beverage for the measurement of glucose, insulin and C-peptide concentrations. Blood glucose concentrations were determined with a glucose analyzer. On Day 28, on which the participant received also investigational product, the OGTT had to be performed prior to consumption of standard meal and administration of investigational product. Unit of measure was millimole × hour per liter)×(milliunits × hour per liter [mmol*h/L)*(mU*h/L]
Measurement of insulin sensitivity consisting of the muscular insulin sensitivity (MISI) obtained during OGTT. | Up to Day 42
  MISI was obtained pre-dose (Day -1), at the end of the dosing period (Day 28), and at end-of-study (Day 42). Blood samples were obtained prior to administration of 75 g of oral glucose which was administered as standard glucose beverage after an overnight fast, within 15 minutes. A peripheral blood sample was drawn from a peripheral arm vein prior to the participant consuming the beverage. Additional blood samples were drawn at 30, 60, 90, and 120 minutes after the participant had consumed the glucose beverage for the measurement of glucose, insulin and C-peptide concentrations. Blood glucose concentrations were determined with a glucose analyzer. On Day 28, on which the participant received also investigational product, the OGTT had to be performed prior to consumption of standard meal and administration of investigational product. Unit of measure was milligram per deciliter per minute per milliunits per liter (mg/dL/min/mU/L).
Measurement of insulin sensitivity consisting of the insulin resistance index obtained during OGTT | Up to Da y 42
  Measurement of insulin sensitivity consisting of the insulin resistance index obtained during OGTT was not collected.
Measurement of insulin sensitivity consisting of the beta cell function based on homeostasis model assessment :HOMA-IR, obtained during OGTT | Up to Day 42
  HOMA-IR was obtained pre-dose (Day -1), at the end of the dosing period (Day 28), and at end-of-study (Day 42). Blood samples were obtained prior to administration of 75 g of oral glucose which was administered as standard glucose beverage after an overnight fast, within 15 minutes. A peripheral blood sample was drawn from a peripheral arm vein prior to the participant consuming the beverage. Additional blood samples were drawn at 30, 60, 90, and 120 minutes after the participant had consumed the glucose beverage for the measurement of glucose, insulin and C-peptide concentrations. Blood glucose concentrations were determined with a glucose analyzer. On Day 28, on which the participant received also investigational product, the OGTT had to be performed prior to consumption of standard meal and administration of investigational product.
Measurement of insulin sensitivity consisting of the beta cell function based on homeostasis model assessment : HOMA-%B, obtained during OGTT. | Up to Day 42
  HOMA-%B was obtained pre-dose (Day -1), at the end of the dosing period (Day 28), and at end-of-study (Day 42). Blood samples were obtained prior to administration of 75 g of oral glucose which was administered as standard glucose beverage after an overnight fast, within 15 minutes. A peripheral blood sample was drawn from a peripheral arm vein prior to the participant consuming the beverage. Additional blood samples were drawn at 30, 60, 90, and 120 minutes after the participant had consumed the glucose beverage for the measurement of glucose, insulin and C-peptide concentrations. Blood glucose concentrations were determined with a glucose analyzer. On Day 28, on which the participant received also investigational product, the OGTT had to be performed prior to consumption of standard meal and administration of investigational product.
Measurement of insulin sensitivity consisting of the quantitative insulin sensitivity check index (QUICKI) obtained during OGTT. | Up to Day 42
  QUICKI was obtained pre-dose (Day -1), at the end of the dosing period (Day 28), and at end-of-study (Day 42). Blood samples were obtained prior to administration of 75 g of oral glucose which was administered as standard glucose beverage after an overnight fast, within 15 minutes. A peripheral blood sample was drawn from a peripheral arm vein prior to the participant consuming the beverage. Additional blood samples were drawn at 30, 60, 90, and 120 minutes after the participant had consumed the glucose beverage for the measurement of glucose, insulin and C-peptide concentrations. Blood glucose concentrations were determined with a glucose analyzer. On Day 28, on which the participant received also investigational product, the OGTT had to be performed prior to consumption of standard meal and administration of investigational product.
Determination of sensitivity and metabolic clearance consisting of the insulin sensitive index (SI), Obtained during an hyperinsulinemic euglycemic glucose clamp (HEGC) | Up to Day 43
  A HEGC was carried out at Day 0, 29 and 43. HEGC was performed in participants who developed coagulation abnormalities during the study. Prior to the start of the HEGC procedure, participants were instructed to refrain from alcohol and caffeine for at least 48 hours before each inpatient visit and from exercise at least 24 hours before each inpatient visit. In the evening of the day prior to the HEGC procedure, the participants received a standard dinner at approximately 19:00 hours. Afterwards, the participants remained fasting until the end of the HEGC procedure at approximately 16:00 hours the next day. The HEGC procedure consisted of three phases: Blood glucose adjustment, Insulin infusion step 1, Insulin infusion step 2. The last 60 min of the two insulin infusion steps were defined as "steady state period 1" (SS1) and "steady state period 2" (SS2). unit of measure was Milliliter per minute permeters squared per micro units (mL/min/m2/mcU/mL).
Determination of insulin sensitivity during first (M1) and second (M2) insulin infusion step. | Up to Day 43
  M1 and M2 was carried out at Day 0, 29 and 43. HEGC was performed in participants who developed coagulation abnormalities during the study. Prior to the start of the HEGC procedure, participants were instructed to refrain from alcohol and caffeine for at least 48 hours before each inpatient visit and from exercise at least 24 hours before each inpatient visit. In the evening of the day prior to the HEGC procedure, the participants received a standard dinner at approximately 19:00 hours. Afterwards, the participants remained fasting until the end of the HEGC procedure at approximately 16:00 hours the next day. The HEGC procedure consisted of three phases: Blood glucose adjustment, Insulin infusion step 1, Insulin infusion step 2. The last 60 min of the two insulin infusion steps were defined as "steady state period 1" (SS1) and "steady state period 2" (SS2). Unit of measure was milligrams per minute per kilograms (mg/min/kg).
Insulin sensitivity in relation to mean insulin infusion concentration (M/I1 and M/I2) ,Obtained during HEGC | Up to Day 43
  M/I1 and M/I2 was carried out at Day 0, 29 and 43. HEGC was performed in participants who developed coagulation abnormalities during the study. Prior to the start of the HEGC procedure, participants were instructed to refrain from alcohol and caffeine for at least 48 hours before each inpatient visit and from exercise at least 24 hours before each inpatient visit. In the evening of the day prior to the HEGC procedure, the participants received a standard dinner at approximately 19:00 hours. Afterwards, the participants remained fasting until the end of the HEGC procedure at approximately 16:00 hours the next day. The HEGC procedure consisted of three phases: Blood glucose adjustment, Insulin infusion step 1, Insulin infusion step 2. The last 60 min of the two insulin infusion steps were defined as "steady state period 1" (SS1) and "steady state period 2" (SS2). milligrams per minute per kilograms per microunits per milliliter (mg/min/kg/μU/mL).
Metabolic clearance rate during first and second insulin infusion step (MCR1, MCR2) on Day 29, and 43 | Up to Day 43
  MCR1, MCR2 was carried out at Day 0, 29 and 43. HEGC was performed in participants who developed coagulation abnormalities during the study. Prior to the start of the HEGC procedure, participants were instructed to refrain from alcohol and caffeine for at least 48 hours before each inpatient visit and from exercise at least 24 hours before each inpatient visit. In the evening of the day prior to the HEGC procedure, the participants received a standard dinner at approximately 19:00 hours. Afterwards, the participants remained fasting until the end of the HEGC procedure at approximately 16:00 hours the next day. The HEGC procedure consisted of three phases: Blood glucose adjustment, Insulin infusion step 1, Insulin infusion step 2. The last 60 min of the two insulin infusion steps were defined as "steady state period 1" (SS1) and "steady state period 2" (SS2). Unit of measure was kilograms per milliliters per kilo calories (kg/mL/kcal)
Variables of metabolic clearance rate including M1ree and M2ree. | Up to Day 43
  M1ree and M2ree was carried out at Day 0, 29 and 43. HEGC was performed in participants who developed coagulation abnormalities during the study. Prior to the start of the HEGC procedure, participants were instructed to refrain from alcohol and caffeine for at least 48 hours before each inpatient visit and from exercise at least 24 hours before each inpatient visit. In the evening of the day prior to the HEGC procedure, the participants received a standard dinner at approximately 19:00 hours. Afterwards, the participants remained fasting until the end of the HEGC procedure at approximately 16:00 hours the next day. The HEGC procedure consisted of three phases: Blood glucose adjustment, Insulin infusion step 1, Insulin infusion step 2. The last 60 min of the two insulin infusion steps were defined as "steady state period 1" (SS1) and "steady state period 2" (SS2).
Variables of metabolic clearance rate including MCR1ree and MCR2ree . | Up to Day 43
  MCR1ree and MCR2ree was carried out at Day 0, 29 and 43. HEGC was performed in participants who developed coagulation abnormalities during the study. Prior to the start of the HEGC procedure, participants were instructed to refrain from alcohol and caffeine for at least 48 hours before each inpatient visit and from exercise at least 24 hours before each inpatient visit. In the evening of the day prior to the HEGC procedure, the participants received a standard dinner at approximately 19:00 hours. Afterwards, the participants remained fasting until the end of the HEGC procedure at approximately 16:00 hours the next day. The HEGC procedure consisted of three phases: Blood glucose adjustment, Insulin infusion step 1, Insulin infusion step 2. The last 60 min of the two insulin infusion steps were defined as "steady state period 1" (SS1) and "steady state period 2" (SS2).
Variables of metabolic clearance rate including M/I1ree and M/I2ree. | Up to Day 43
  M/I1ree and M/I2ree was carried out at Day 0, 29 and 43. HEGC was performed in participants who developed coagulation abnormalities during the study. Prior to the start of the HEGC procedure, participants were instructed to refrain from alcohol and caffeine for at least 48 hours before each inpatient visit and from exercise at least 24 hours before each inpatient visit. In the evening of the day prior to the HEGC procedure, the participants received a standard dinner at approximately 19:00 hours. Afterwards, the participants remained fasting until the end of the HEGC procedure at approximately 16:00 hours the next day. The HEGC procedure consisted of three phases: Blood glucose adjustment, Insulin infusion step 1, Insulin infusion step 2. The last 60 min of the two insulin infusion steps were defined as "steady state period 1" (SS1) and "steady state period 2" (SS2).
Mean steady state concentration Free fatty acids (FFA), and glycerols | Up to Day 43
  Mean steady state concentration Free fatty acids and glycerols was carried out at Day 0, 29 and 43. HEGC was performed in participants who developed coagulation abnormalities during the study. Prior to the start of the HEGC procedure, participants were instructed to refrain from alcohol and caffeine for at least 48 hours before each inpatient visit and from exercise at least 24 hours before each inpatient visit. In the evening of the day prior to the HEGC procedure, the participants received a standard dinner at approximately 19:00 hours. Afterwards, the participants remained fasting until the end of the HEGC procedure at approximately 16:00 hours the next day. The HEGC procedure consisted of three phases: Blood glucose adjustment, Insulin infusion step 1, Insulin infusion step 2. The last 60 min of the two insulin infusion steps were defined as "steady state period 1" (SS1) and "steady state period 2" (SS2).
Mean C-peptide concentration (mean C-peptideSS1 and C-peptideSS2) obtained during HEGC | Up to Day 43
  Mean C-peptideSS1 and C-peptideSS2 was carried out at Day 0, 29 and 43. HEGC was performed in participants who developed coagulation abnormalities during the study. Prior to the start of the HEGC procedure, participants were instructed to refrain from alcohol and caffeine for at least 48 hours before each inpatient visit and from exercise at least 24 hours before each inpatient visit. In the evening of the day prior to the HEGC procedure, the participants received a standard dinner at approximately 19:00 hours. Afterwards, the participants remained fasting until the end of the HEGC procedure at approximately 16:00 hours the next day. The HEGC procedure consisted of three phases: Blood glucose adjustment, Insulin infusion step 1, Insulin infusion step 2. The last 60 min of the two insulin infusion steps were defined as "steady state period 1" (SS1) and "steady state period 2" (SS2).
Number of participants with all adverse events (AEs) and serious adverse events (SAEs) | Up to 28 days
  Data for number of participants who presented one or more adverse events (serious or non serious) was reported. An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Number of participants with hypoglycemic events | Up to Day 28
  Symptomatic, symptomatic and Severe Symptomatic hypoglycemia definitions were used to analyze and report hypoglycemic events. Symptomatic hypoglycemic episodes were collected from Day 1 to Day 28 with the assistance of participants diaries. Symptomatic hypoglycemia and severe symptomatic hypoglycemia was recorded in CRFs as AEs in all cases.
Number of participants with abnormal Physical examination findings | Up to Day 41
  A complete physical examination, including an ophthalmological examination to rule out diabetic neuropathy, was performed at screening. A symptom-driven, directed physical examination was performed also pre dosing (Day-2), during the dosing period (Day 14 and 27) and after dosing (Day 41). Number of participants with abnormal physical findings was reported.
Change from baseline in Vital signs-systolic blood pressure (SBP) and diastolic blood pressure (DBP). | Up to Day 43
  SBP and DBP were investigated at screening, pre-dosing (Day -2), during the dosing period (Day 1, 14 and 27) and at end of dosing follow-up period/end-of-study (Day 41 and 43).
  At Day 1 the vital signs were collected pre-dose (baseline values) and 3 hours post-dose. Day 0 was Baseline and change from Baseline was a value at study day subtracted by value at baseline.
Change from baseline in Vital signs-Heart rate | Up to Day 43
  Heart rate was investigated at screening, pre-dosing (Day -2), during the dosing period (Day 1, 14 and 27) and at end of dosing follow-up period/end-of-study (Day 41 and 43). At Day 1 the vital signs were collected pre-dose (baseline values) and 3 hours post-dose. Day 0 was Baseline and change from Baseline was a value at study day subtracted by value at baseline.
Change from baseline in Vital signs-Respiratory rate | Up to Day 43
  Respiratory rate was investigated at screening, pre-dosing (Day -2), during the dosing period (Day 1, 14 and 27) and at end of dosing follow-up period/end-of-study (Day 41 and 43). At Day 1 the vital signs were collected pre-dose (baseline values) and 3 hours post-dose. Day 0 was Baseline and change from Baseline was a value at study day subtracted by value at baseline.
Change from baseline in Vital signs-Temperature. | Up to Day 43
Number of participants with abnormal electrocardiogram (ECG) recordings | Up to Day 43
  A 12-lead ECG was recorded at screening, pre-dose (Day -2), at the beginning and end of the dosing period (Day 1 and 27) and at the end of the dosing follow-up period/end-of study (Day 41 and 43). Number of participants with abnormal ECG findings was reported.
Mean hematology parameters including white blood cell (WBC) and platelets count | Up to Day 42
  Blood samples for assessment of WBC and platelet count was collected at screening, Day -1, 14, 28 and 42. Data for mean and standard deviation was presented.
Mean hematology parameters including WBC Differential count and Red cell distribution width (RDW) | Up to Day 42
  Blood samples for assessment of WBC differential count and RDW was collected at screening, Day -1, 14, 28 and 42. Data for mean and standard deviation was presented.
Mean hematology parameters including Hemoglobin (Hb) and Mean corpuscular hemoglobin concentration (MCHC) | Up to Day 42
  Blood samples for assessment of Hb and MCHC was collected at screening, Day -1, 14, 28 and 42. Data for mean and standard deviation was presented.
Mean hematology parameters including: hematocrit count | Up to Day 42
  Blood samples for assessment of hematocrit count was collected at screening, Day -1, 14, 28 and 42. Data for mean and standard deviation was presented.
Mean hematology parameters including corpuscular volume (MCV) | Up to Day 42
  Blood samples for assessment of MCV was collected at screening, Day -1, 14, 28 and 42. Data for mean and standard deviation was presented.
Mean hematology parameters including corpuscular hemoglobin (MCH) | Up to Day 42
  Blood samples for assessment of MCH was collected at screening, Day -1, 14, 28 and 42. Data for mean and standard deviation was presented.
Mean hematology parameters including Red Blood Cells (RBCs) count | Up to Day 42
  Blood samples for assessment of RBC count was collected at screening, Day -1, 14, 28 and 42. Data for mean and standard deviation was presented.
Summary of urinalysis data: PH | Up to Day 42
  Samples for pH assessment were collected at screening, Day -1, 14, 28 and 42. Unscheduled and control assessments were not included in the analysis. Data for mean and standard deviation was presented.
Number of participants with urinalysis | Up to Day 42
  Data for urinalysis was collected at screening, Day -1, 14, 28 and 42. Data for participants with positive and negative urinalysis result was presented. Unscheduled and control assessments were not included in the analysis.
Mean clinical chemistry parameters including calcium, chloride, magnesium, potassium, sodium, bicarbonate, phosphate, glucose, urea and blood urea | Up to Day 42
  Clinical chemistry assessment for calcium, chloride, magnesium, potassium, sodium, bicarbonate, phosphate, glucose, urea ,blood urea was done at screening, Day -1, 14, 28 and 42. Data for mean and standard deviation was presented.
Mean clinical chemistry parameters including direct bilirubin, indirect bilirubin, total bilirubin ,uric acid | Up to Day 42
  Clinical chemistry assessment for direct bilirubin, indirect bilirubin, total bilirubin and uric acid was done at screening, Day -1, 14, 28 and 42. Data for mean and standard deviation was presented.
Mean clinical chemistry parameters including alkaline phosphatase (ALP), Alanine aminotransferase (ALT), Aspartate aminotransaminase (AST), Lactate dehydrogenase (LDH), Creatine kinase | Up to Day 42
  Clinical chemistry assessment for ALP, ALT, AST, LDH and creatine kinase was done at screening, Day -1, 14, 28 and 42. Data for mean and standard deviation was presented.
Mean clinical chemistry parameters including albumin | Up to Day 42
  Clinical chemistry assessment for albumin was done at screening, Day -1, 14, 28 and 42. Data for mean and standard deviation was presented.
Mean clinical chemistry parameters including serum creatinine | Up to Day 42
  Clinical chemistry assessment for serum creatinine was done at screening, Day -1, 14, 28 and 42. Data for mean and standard deviation was presented.

SECONDARY OUTCOMES:
The area under the plasma concentration time curve of SRT2104 from time 0 (dosing) to 24 hours post-dose (AUC 0-24h) | Day 1 and 28 at pre-dose, and at 15, 30 minutes,1, 2, 3, 4, 8, 12 and 24 hours
  Approximately 90 mL of blood was collected throughout duration of the trial for determination of SRT2104 in plasma. Samples were collected on Days 1 and 28 at pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours and for analysis. Blood samples were drawn via an indwelling cannula on days with multiple samples. unit of measure was nanograms × hours per milliliter ( ng*h/mL)
The area under the plasma concentration time curve of SRT2104 from time 0 to infinity (AUC 0-∞) | Day 1 and 28 at pre-dose, and at 15, 30 minutes,1, 2, 3, 4, 8, 12 and 24 hours
  The AUC (from zero to infinity) represents the total drug exposure over time. Approximately 90 mL of blood was collected throughout duration of the trial for determination of SRT2104 in plasma. Samples were collected on Days 1 and 28 at pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours and for analysis. Blood samples were drawn via an indwelling cannula on days with multiple samples.
Mean maximum plasma concentration of SRT2104 (Cmax) | Day 1 and 28 at pre-dose, and at 15, 30 minutes,1, 2, 3, 4, 8, 12 and 24 hours
  Cmax refers to the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and before the administration of a second dose. Approximately 90 mL of blood was collected throughout duration of the trial for determination of SRT2104 in plasma. Samples were collected on Days 1 and 28 at pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours and for analysis. Blood samples were drawn via an indwelling cannula on days with multiple samples.
Mean time to maximum plasma SRT2104 concentration (tmax) | Day 1 and 28 at pre-dose, and at 15, 30 minutes,1, 2, 3, 4, 8, 12 and 24 hoursDay 1, 2, 28, and 29
  tmax is the term used in pharmacokinetics to describe the time at which the Cmax is observed Approximately 90 mL of blood was collected throughout duration of the trial for determination of SRT2104 in plasma. Samples were collected on Days 1 and 28 at pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours and for analysis. Blood samples were drawn via an indwelling cannula on days with multiple samples.
Mean Terminal elimination rate constant of SRT2104 (ƛz) | Day 1 and 28 at pre-dose, and at 15, 30 minutes,1, 2, 3, 4, 8, 12 and 24 hours
  Approximately 90 mL of blood was collected throughout duration of the trial for determination of SRT2104 in plasma. Samples were collected on Days 1 and 28 at pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours and for analysis. Blood samples were drawn via an indwelling cannula on days with multiple samples.
Mean terminal plasma elimination half time (t1/2) of SRT2104. | Day 1 and 28 at pre-dose, and at 15, 30 minutes,1, 2, 3, 4, 8, 12 and 24 hours
  terminal plasma elimination half time (t1/2) was derived from plasma concentration versus time data. (t1/2) was the time required for one half of the total amount of administered drug to be eliminated from the body. Approximately 90 mL of blood was collected throughout duration of the trial for determination of SRT2104 in plasma. Samples were collected on Days 1 and 28 at pre-dose and at 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours and for analysis. Blood samples were drawn via an indwelling cannula on days with multiple samples.
Energy expenditure (indirect calorimetry) parameters-Oxygen consumption (% O2) at ss1 and ss2 | Up to Day 43
  Oxygen consumption was reported using indirect calorimetry. Indirect calorimetry was performed using Quark RMR (COSMED, Rome, Italy) on Day 0, 29 and 43 during the HEGC procedure for four 30-minute sessions at time points -570 min to -540 min (baseline), -40 min to -10 min (end of blood glucose adjustment phase), 210 min to 240 min (end of SS1), 450 min to 480 min (end of SS2).
Energy expenditure (indirect calorimetry) parameters- Carbon dioxide production(CO2) at ss1 and ss2 | Up to Day 43
  Carbon dioxide production was reported using indirect calorimetry. Indirect calorimetry was performed using Quark RMR (COSMED, Rome, Italy) on Day 0, 29 and 43 during the HEGC procedure for four 30-minute sessions at time points -570 min to -540 min (baseline), -40 min to -10 min (end of blood glucose adjustment phase), 210 min to 240 min (end of SS1), 450 min to 480 min (end of SS2).
Energy expenditure (indirect calorimetry) parameters-Resting energy expenditure (ree) at ss1 and ss2 | Up to Day 43
  Resting energy expenditure was reported using indirect calorimetry. Indirect calorimetry was performed using Quark RMR (COSMED, Rome, Italy) on Day 0, 29 and 43 during the HEGC procedure for four 30-minute sessions at time points -570 min to -540 min (baseline), -40 min to -10 min (end of blood glucose adjustment phase), 210 min to 240 min (end of SS1), 450 min to 480 min (end of SS2).
Energy expenditure (indirect calorimetry) parameters Carbohydrate/glucose oxidation rate (c) at ss1 and ss2 | Up to Week 43
  Carbohydrate/glucose oxidation rate was reported using indirect calorimetry. Indirect calorimetry was performed using Quark RMR (COSMED, Rome, Italy) on Day 0, 29 and 43 during the HEGC procedure for four 30-minute sessions at time points -570 min to -540 min (baseline), -40 min to -10 min (end of blood glucose adjustment phase), 210 min to 240 min (end of SS1), 450 min to 480 min (end of SS2).
Energy expenditure (indirect calorimetry) parameters- Fat oxidation rate (f) at ss1 and ss2 | up to Day 43
  Fat oxidation rate was reported using indirect calorimetry. Indirect calorimetry was performed using Quark RMR (COSMED, Rome, Italy) on Day 0, 29 and 43 during the HEGC procedure for four 30-minute sessions at time points -570 min to -540 min (baseline), -40 min to -10 min (end of blood glucose adjustment phase), 210 min to 240 min (end of SS1), 450 min to 480 min (end of SS2).
Energy expenditure (indirect calorimetry) parameters-Urinary urea excretion rate (n) | Up to Day 43
  Urinary urea excretion rate was reported using indirect calorimetry. Indirect calorimetry was performed using Quark RMR (COSMED, Rome, Italy) on Day 0, 29 and 43 during the HEGC procedure for four 30-minute sessions at time points -570 min to -540 min (baseline), -40 min to -10 min (end of blood glucose adjustment phase), 210 min to 240 min (end of SS1), 450 min to 480 min (end of SS2).
Energy expenditure (indirect calorimetry) parameters-Oxidative and non- oxidative glucose disposal (VO2 and VCO2) at ss1 and ss2 | Up to Day 43
  Oxidative and non- oxidative glucose disposal was reported using indirect calorimetry. Indirect calorimetry was performed using Quark RMR (COSMED, Rome, Italy) on Day 0, 29 and 43 during the HEGC procedure for four 30-minute sessions at time points -570 min to -540 min (baseline), -40 min to -10 min (end of blood glucose adjustment phase), 210 min to 240 min (end of SS1), 450 min to 480 min (end of SS2).
Energy expenditure (indirect calorimetry )parameters-Respiratory exchange ratio (RER) | Up to Day 43
  RER was defined as the ratio between the amount of O2 consumed and CO2 produced in one breath. The parameter was assessed during indirect measure of heat production (calorimetry).
Mean 7-point-blood glucose-AUC | Up to Day 42
  AUC was presented using a 7-point blood glucose profile was performed during the inpatient portion of the study (Day -1, 28 and 42) to measure and record glucose levels throughout the day. Blood glucose concentrations were determined with a glucose analyzer. The first sample was collected early in the morning before the OGTT and standardized meal.
Muscle histology and biomarkers of oxidative capacity -mitochondrial deoxyribonucleic acid (DNA). | Up to Day 28
  Muscle biopsies were obtained pre-dose (Day -1) and at end of the dosing period (Day 28)
Muscle histology and biomarkers of oxidative capacity-Citrase synthase activity (Complex I) | Up to Days 28
  Muscle biopsies were obtained pre-dose (Day -1) and at end of the dosing period (Day 28) Data for mean and standard deviation was presented.
Muscle histology and biomarkers of oxidative capacity-Citrase synthase activity (Complex II/III and IV) | Up to Day 28
  Muscle biopsies were obtained pre-dose (Day -1) and at end of the dosing period (Day 28) Data for mean and standard deviation was presented.
Muscle histology and biomarkers of oxidative capacity-succinate dehydrogenase content Complex I, Complex II/III, complex IV. | Day 0, 29, and 43
  Muscle biopsies were obtained pre-dose (Day -1) and at end of the dosing period (Day 28) Data for mean and standard deviation was presented.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register